CLINICAL TRIAL: NCT06552130
Title: The Importance of Insulin Action in the Brain for the Immune System During Physical Activity
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ulm (Other)
Responsible Party: Principal Investigator, Martin Heni, Head of the Section Endocrinology and Diabetology, Full Professorship (W3) for Endocrinology and Diabetology, University of Ulm
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 81/24
Record Dates: First submitted 2024-08-02; First posted 2024-08-13 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Insulin Sensitivity
Keywords: brain insulin action; autonomic nervous system; physical activity
MeSH Terms: conditions — Insulin Resistance; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intranasal insulin spray (Experimental): 160 Units of human insulin as nasal spray
  Interventions: Other: Spiroergometer test with intranasal insulin spray
- Placebo spray (Placebo Comparator): Nasal spray containing placebo solution
  Interventions: Other: Spiroergometer test with intranasal placebo spray

INTERVENTIONS:
Other: Spiroergometer test with intranasal insulin spray — Participants will undergo a 60 min bicycle spiroergometer test and intranasal insulin spray. Intranasal insulin will be administered 30 minutes prior to the start of the physical activity.
  Arms: Intranasal insulin spray
Other: Spiroergometer test with intranasal placebo spray — Participants will undergo a 30 min bicycle spiroergometer test and intranasal placebo spray. To mimic insulin spill-over from nasal spray into systemic circulation, an i.v. insulin bolus of 3 mU × kg-1. will be administered over 15 minutes 30 minutes prior to the start of the physical activity on the placebo spray day. On the insulin spray day a comparable amount of saline will be infused.
  Arms: Placebo spray

SUMMARY:
The goal of this clinical trial is to clarify the interaction of central insulin action and physical activity with the immune system.

Therefore, participants will undergo bicycle spiroergometer tests. This approach will be compared between days with insulin delivery to the brain as nasal spray and days with placebo spray.

DETAILED DESCRIPTION:
This research project aims to investigate if the brain insulin action regulates the immune system via the autonomous nervous system during physical activity.

Therefore, insulin action in the brain will be introduced by application of insulin as nasal spray (on one day) versus carrier solution as placebo nasal spray (on another day) in a randomized, blinded fashion. Spray administration will be performed 30 minutes before a 60 min bicycle spiroergometer test at 70 % VO2max that will introduce a postprandial state. On placebo day, the known spillover of tiny amounts of nasal insulin into the systemic circulation will be mimicked by an appropriate i.v. insulin bolus. Using this approach, brain-derived regulation of the immune system including the stimulation of immune cells via cytokines, physical performance, activity of the autonomous nervous system and gene-expression of leukocytes will be examined.

ELIGIBILITY:
Inclusion Criteria:

* BMI < 24 kg/m2
* no known primary diseases
* hormonal contraception with a single-phase preparation

Exclusion Criteria:

* Alcohol or drug abuse
* Smoking
* At screening: Hb < 12 g/dl for women and Hb < 14 g/dl for men
* Any (clinical) condition that would endanger participant's safety or question scientific success according to a physician's opinion.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2024-12-15 (Actual); Primary Completion 2025-08-14 (Actual); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Immune system activation | 120 minutes
  Influence of central nervous insulin action on the activation of the immune system activation by exercise, measured by circulating cytokines and cytokines in the supernatant of stimulated peripheral blood mononuclear cells.
Immune system activation | 120 minutes
  Influence of central nervous insulin action on the activation of the immune system activation by exercise, measured by the composition of immune cells in circulation and cytokine release in the supernatant of stimulated peripheral blood mononuclear cells.

SECONDARY OUTCOMES:
Maximal oxygen consumption (VO2max) | 60 minutes
  Influence of central nervous insulin action on physical performance measured as VO2 peak during spiroergometry.
Heart rate variability | 120 minutes
  Influence of central nervous insulin action on the activity of the autonomic nervous system recorded by means of heart rate variability from an electrocardiogram.
Corticotropic pituitary axis modulation | 120 minutes
  Influence of central nervous insulin action in the activity of the corticotropin pituitary axis during physical activity, measured by cortisol, dehydroepiandrosterone and adrenocorticotropic hormone
Leukocyte gene expression | 120 minutes
  Influence of central nervous insulin action on the gene expression of leukocytes during physical activity
Individual anaerobic threshold | 120 minutes
  Influence of central nervous insulin action on physical performance. Individual anaerobic threshold assessed by lactate measurement from venous blood sampling.
Catecholamines | 120 minutes
  Influence of central nervous insulin action on the activity of the autonomic nervous system recorded by means of measuring catecholamine concentrations from venous blood.
Effects on blood coagulation parameters | 120 Minutes
  Influence of central nervous insulin action and/or physical activity on blood coagulation parameters assessed through global coagulation tests and single coagulation factors.

OTHER OUTCOMES:
sex differences | 120 minutes
  Potential differences in the above mentioned outcomes between sexes will be analyzed.

CONTACTS AND LOCATIONS:
Overall Officials: Martin Heni, MD, Principal Investigator — University of Ulm
Locations (1):
- Universityhospital Ulm, Ulm, Germany